CLINICAL TRIAL: NCT01788020
Title: Efficacy of First Line Dexamethasone, Rituximab and Cyclophosphamide (DRC) +/- Bortezomib for Patients With Waldenström's Macroglobulinemia
Brief Title: Efficacy of First Line DRC +/- Bortezomib for Patients With Waldenström's Macroglobulinemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Centre Hospitalier de Lens (Co-Sponsor) (Unknown)
Responsible Party: Principal Investigator, Christian Buske, Prof. Dr. med. Christian Buske, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECWM-1; 2013-000506-37 (EudraCT Number)
Record Dates: First submitted 2013-02-01; First posted 2013-02-11 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Waldenström's Macroglobulinemia
Keywords: DRC; Bortezomib; Oncology
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Neoplasms | interventions — Dexamethasone; Rituximab; Cyclophosphamide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DRC+Bortezomib (Experimental): Induction experimental arm (Arm B):
  Cycle 1:
  Bortezomib 1.6 mg/m2 s.c. Day 1,8,15; Dexamethasone 20 mg p.o. Day 1; Rituximab 375 mg/m2 i.v. Day 1; Cyclophosphamide 100 mg/m2 x 2 p.o. Day 1-5
  Cycle 2-6:
  Bortezomib 1.6 mg/m2 s.c. Day 1,8,15; Dexamethasone 20 mg p.o. Day 1; Rituximab 1400 mg absolute sc Day 1; Cyclophosphamide 100 mg/m2 x 2 p.o. Day 1-5; Repeat day 29.
  Interventions: Drug: Dexamethasone, Rituximab, Cyclophosphamide, Bortezomib
- DRC (Active Comparator): Induction standard arm (Arm A)
  Cycle 1:
  Dexamethasone 20 mg p.o. Day 1; Rituximab 375 mg/m2 i.v. Day 1; Cyclophosphamide 100 mg/m2 x 2 p.o. Day 1-5;
  Cycle 2-6:
  Dexamethasone 20 mg p.o. Day 1; Rituximab 1400 mg absolute sc Day 1; Cyclophosphamide 100 mg/m2 x 2 p.o. Day 1-5; Repeat day 29.
  Interventions: Drug: Dexamethasone, Rituximab, Cyclophosphamide

INTERVENTIONS:
Drug: Dexamethasone, Rituximab, Cyclophosphamide
  Arms: DRC
Drug: Dexamethasone, Rituximab, Cyclophosphamide, Bortezomib
  Arms: DRC+Bortezomib

SUMMARY:
In Waldenström macroglobulinemia (WM) conventional chemotherapy induces only low CR rates and responses of short duration compared to other indolent lymphomas. Thus innovative approaches are needed which combine excellent activity and tolerability in patients with WM, who are mostly of advanced age. The immunochemotherapy DRC (dexamethasone, rituximab, cyclophosphamide) was shown to be highly effective in patients with WM without inducing major hematological toxicities. On the other hand the proteasome inhibitor Bortezomib showed substantial activity as a single agent in WM with only very few side effects when given in a weekly schedule. Based on these observations it is the aim of this study to test whether the efficacy of the well tolerated DRC regime can be further improved by adding Bortezomib.

DETAILED DESCRIPTION:
Waldenström's macroglobulinemia (WM) is defined by a bone marrow infiltration by lymphoplasmacytic cells and the presence of a monoclonal immunoglobulin (Ig) M gammopathy in the peripheral blood. The clinical understanding of the disease has been greatly improved by the identification of internationally recognized criteria for initiating therapy, the description of an international prognostic index for patients requiring a first-line therapy and the definition of response criteria. These criteria are mainly based on the evolution of serum IgM concentration. However, delayed IgM monoclonal protein responses may cause important difficulties in response assessment. In addition, discrepancies between the kinetics of serum M protein reduction and the clearance of monoclonal B-cells from the bone marrow have been reported. Despite continuing advances in the therapy of WM, the disease remains incurable with a median survival of 5 to 8 years from the time of diagnosis thereby necessitating the development and evaluation of novel treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

Clinicopathological diagnosis of WM as defined by consensus panel one of the Second International Workshop on WM. Pathological diagnosis has to occur before study inclusion and randomization. In addition, pathological specimens have to be sent to the national pathological reference center at study inclusion and randomization. The positivity for CD20 can be assumed from any previous bone marrow immunohistochemistry or flow cytometry analysis performed up to 6 months prior to enrollment. Inclusion in the study will be based on morphological and immunological criteria. Immunophenotyping will be performed in each center and saved locally. Flow cytometry of bone marrow and blood cells will include at least one double staining and assess the expression of the following antigens: surface immunoglobulin, CD19, CD20, CD5, CD10 and CD23. Patients are eligible if tumor cells express the following antigens: CD19, CD20, and if they are negative for CD5, CD10 and CD23 expression. Patients with tumor cells positive for CD5 and/or CD23 and morphologically similar to WM cells may be included after ruling out other low grade B-cell malignancies.

* Presence of at least one criterion for initiation of therapy, according to the 2nd Workshop on WM:

  * Recurrent fever, night sweats, weight loss, fatigue
  * Hyperviscosity
  * Lymphadenopathy which is either symptomatic or bulky (≥5 cm in maximum diameter)
  * Symptomatic hepatomegaly and/or splenomegaly
  * Symptomatic organomegaly and/or organ or tissue infiltration
  * Peripheral neuropathy due to WM
  * Symptomatic cryoglobulinemia
  * Cold agglutinin anemia
  * IgM related immune hemolytic anemia and/or thrombocytopenia
  * Nephropathy related to WM
  * Amyloidosis related to WM
  * Hemoglobin ≤10g/dL
  * Platelet count <100x10^9/L
  * Serum monoclonal protein >5g/dL, even with no overt clinical symptoms Cumulative illness rating scale (CIRS) score less than 6
* World Health Organization (WHO)/ECOG performance status 0 to 2.
* Other criteria:

  * Age ≥ than 18 years
  * Life expectancy >3 months.
  * Baseline platelet count ≥ 50 ×10^9/L, absolute neutrophil count ≥ 0.75×10^9/L (if not due to BM infiltration by the lymphoma).
  * Meet the following pretreatment laboratory criteria at the Screening visit conducted within 28 days of study enrollment:

    * ASAT (SGOT): ≤3 times the upper limit of institutional laboratory normal value
    * ALAT (SGPT): ≤3 times the upper limit of institutional laboratory normal value
    * Total Bilirubin: ≤20 mg/L or 2 times the upper limit of institutional laboratory normal value, unless clearly related to the disease (except if due to Gilbert's syndrome)
    * Serum creatinine: ≤ 2mg/dl
* Premenopausal fertile females must agree to use a highly effective method of birth control for the duration of the therapy up to 6 months after end of therapy. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
* Men must agree not to father a child for the duration of therapy and 6 months after and must agree to advice a female partner to use a highly effective method of birth control.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion criteria:

* Prior systemic treatment of the WM (plasmapheresis and short- term administration of corticosteroids < 4 weeks administered at a dose equivalent to < 20 mg/day prednisone is allowed)
* Patient with hypersensitivity to dexamethasone.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Uncontrolled bacterial, viral or fungal infection
* Active HIV, HBV or HCV infection
* Known interstitial lung disease
* Prior allergic reaction or severe anaphylactic reaction related to humanized or murine monoclonal antibody.
* Central Nervous System involvement by lymphoma
* Prior history of malignancies unless the subject has been free of the disease for ≥ 5 years. Exceptions include the following:

  * Basal cell carcinoma of the skin,
  * Squamous cell carcinoma of the skin,
  * Carcinoma in situ of the cervix,
  * Carcinoma in situ of the breast,
  * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b).
* Uncontrolled illness including, but not limited to:

  * Uncontrolled diabetes mellitus mellitus (as indicated by metabolic derangements and/or severe diabetes mellitus related uncontrolled organ complications)
  * Chronic symptomatic congestive heart failure (Class NYHA III or IV).
  * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
  * Clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia.
  * Known pericardial disease
* Subjects with ≥ Grade 2 neuropathy.
* Women who are pregnant as well as women who are breastfeeding and do not consent to discontinue breast-feeding.
* Participation in another clinical trial within four weeks before randomization in this study
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician about study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-11; Primary Completion 2018-11 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | participants will be followed for their participation in the trial, an expected average of 5.5 years
  PFS will be calculated from the date of inclusion/randomisation to the following events: the date of progression and the date of death if it occurred earlier. In the absence of progression and death, PFS duration will be censored at the stopping date or the date of last follow-up.

SECONDARY OUTCOMES:
Response rate | 24 weeks
  The response rates (CR,VGPR, PR, MR) and overall response rate (CR, VGPR, PR, MR) are evaluated 4 weeks after the end of induction treatment.
Best response | 24 weeks
  Best response is determined in the time interval from the start of induction therapy to end of follow-up.
Time to best response | 24 weeks
  Time to best response is defined as the time from the start of induction to best response the patient achieves (CR, VGPR, PR, MR).
Time to first response | 24 weeks
  Time to first response is defined as the time from the start of induction to first response (MR, PR, VGPR or CR).
Time to treatment failure | participants will be followed for their participation in the trial, an expected average of 5.5 years
  Time to treatment failure (TTF) is defined as the time of randomization to discontinuation of therapy for any reason including death from any cause, progression, toxicity or add-on of new anti-cancer therapy. Patients alive without treatment failure are censored at the latest tumor assessment date.
Remission duration | participants will be followed for their participation in the trial (from date of response), an expected average of 5 years
  Remission duration will be calculated in patients with response (CR, VGPR, PR, MR) to induction from end of induction to the date of progression, relapse or death from any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
Cause specific survival (CSS) | participants will be followed for their participation in the trial, an expected average of 5.5 years
  Cause specific survival is defined as the period from the induction randomization to death from lymphoma or lymphoma related cause; death unrelated to WM is considered as a competing event.
Overall survival (OS) | participants will be followed for their participation in the trial, an expected average of 5.5 years]
  Overall survival is defined as the period from the induction randomization to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dreyling, MD, Principal Investigator — National Co-Coordinating Investigator - Germany University Hospital Großhadern, Munich; Veronique Leblond, MD, Principal Investigator — National Co-Coordinating Investigator - Groupe Hospitalier Pitié Salpêtrière France (Paris); Pierre Morel, MD, Principal Investigator — National Co-Coordinating Investigator - Centre Hospitalier Schaffner France (Lens cedex); Garcia Sanz, MD, Principal Investigator — National Co-Coordinating Investigator - University Hospital Salamanca Spain; Maria da Silva, MD, Principal Investigator — National Co-Coordinating Investigator - Portuguese Institute of Oncology Portugal; Meletios Dimopoulos, MD, Principal Investigator — National Co-Coordinating Investigator - University of Athens School of Medicine Athens Greece; Eva Kimby, MD, Principal Investigator — National Co-Coordinating Investigator - Sweden, Denmark, Norway Hematology and Internal Medicine Karolinska Institutet Stockholm Sweden; Roman Hajek, MD, Principal Investigator — National Co-Coordinating Investigator - Department of Haematooncology Ostrava Czech Republic; Wolfram Klapper, MD, Study Chair — Coordinator Pathology (Germany) Department of Pathology Kiel; Sylvie Chevret, Study Chair — Central Statistics (France)Department of Biostatistics and Medical Information,Hôpital Saint Louis, Paris; Christian Buske, MD, Study Director — Coordinating Investigator Germany University Hospital Ulm
Locations (1):
- University Hospital Ulm, Ulm, Germany

REFERENCES:
- [Background] Buske C, Dimopoulos MA, Grunenberg A, Kastritis E, Tomowiak C, Mahe B, Troussard X, Hajek R, Viardot A, Tournilhac O, Aurran T, Lepretre S, Zerazhi H, Hivert B, Leblond V, de Guibert S, Brandefors L, Garcia-Sanz R, Gomes da Silva M, Kimby E, Schmelzle B, Kaszynski D, Dreyhaupt J, Muche R, Morel P. Bortezomib-Dexamethasone, Rituximab, and Cyclophosphamide as First-Line Treatment for Waldenstrom's Macroglobulinemia: A Prospectively Randomized Trial of the European Consortium for Waldenstrom's Macroglobulinemia. J Clin Oncol. 2023 May 10;41(14):2607-2616. doi: 10.1200/JCO.22.01805. Epub 2023 Feb 10. PMID 36763945